CLINICAL TRIAL: NCT02193620
Title: A Randomized, Double Blind, Placebo-controlled, Multiple Dose Study to Assess the Efficacy, Safety and Pharmacokinetics of Oral Nalbuphine, an Oral Soft Capsule, for Post-hemorrhoidectomy Pain Management
Brief Title: Study of PHN131 in Patients After Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PH-CP025
Record Dates: First submitted 2014-07-14; First posted 2014-07-17 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Analgesia Disorder
Keywords: Analgesic; Narcotics; Opioids; Pain relief after surgery
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): Placebo soft capsules
  Interventions: Drug: Placebo soft capsules; Drug: Dicofenac
- Study group (Experimental): PHN131 soft capsule with Nalbuphine HCl 60 mg/cap
  Interventions: Drug: PHN131 soft capsule with Nalbuphine HCl 60 mg/cap; Drug: Dicofenac

INTERVENTIONS:
Drug: PHN131 soft capsule with Nalbuphine HCl 60 mg/cap — Multiple dose of oral PHN131 soft capsule with Nalbuphine HCl 60 mg/cap, initial dose : 120 mg ( 2 capsules), then 60 mg (1 capsule); t.i.d.
  Other Names: PHN131
  Arms: Study group
Drug: Placebo soft capsules — Multiple dose of oral Placebo soft capsules, initial dose: 2 capsules, then 1 capsule; t.i.d.
  Other Names: Placebo
  Arms: Placebo group
Drug: Dicofenac — All subjects will receive diclofenac by IM injection for analgesia as rescue pain control.

SUMMARY:
The purpose of this study is to assess the effectiveness, safety and pharmacokinetics of Oral Nalbuphine in the treatment of postoperative pain following hemorrhoidectomy.

DETAILED DESCRIPTION:
• Primary Efficacy Endpoint: Pain assessment calculated as the area under the curve of VAS pain intensity scores through 48 hours.

• Secondary Efficacy Endpoints:

1. Consumption of diclofenac (Day 1-2) via Intramuscular Injection (IM injection).
2. Time from the end of operation to the first IM injection diclofenac dose
3. Brief Pain Inventory (BPI).
4. Patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >= 20 years of age at Screening
2. Scheduled to electively undergo 2 or 3-column excisional hemorrhoidectomy
3. American Society of Anesthesiology Physical Class 1 - 3
4. Clinical lab values twice the upper limit of normal (values of potential clinical concern are detailed in Appendix) or, if abnormal, deemed not clinically significant per the Investigator.
5. Ability and willingness to provide informed consent, adhere to the study visit schedule and complete all study assessments and language specific questionnaires.

Exclusion Criteria:

1. Body weight less than 40 kg.
2. Concurrent fissurectomy.
3. Subject is pregnant or breastfeeding. Women of childbearing potential must have a negative urine pregnancy test at Baseline.
4. Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study.
5. History of hypersensitivity or allergy to amide-type local anesthetics, opioid, or any ingredient of the medications administered in this study.
6. Subject has a resting respiratory rate less than 8 per minute and blood oxygen saturation less than 90 mmHg.
7. Use of any NSAIDs, selective COX-2 inhibitors, opioid, acetaminophen, selective serotonin reuptake inhibitors (SSRI), tricyclic antidepressants (TCA), gabapentin, or pregabalin within three days of surgery.
8. Chronic use of opioid medications for more than 14 days in the last 3 months, or non-opioid pain medications more than 5 times per week.
9. Use of any long-acting opioid medication within 3 days of surgery or any opioid medication within 24 hours of surgery.
10. Current painful physical condition or concurrent surgery requires analgesic treatment in the postoperative period.
11. Contraindication to epinephrine or any of the pain-control agents planned for postoperative use.
12. Administration of an investigational drug within the longer of 30 days or 5 elimination half-lives of such investigational drug prior to study drug administration.
13. Any psychiatric disorder, psychological, medical, or laboratory condition that may interfere with study assessments or compliance.
14. Significant medical conditions or laboratory results that may indicate an increased vulnerability to study drugs and procedures, and thus expose the subject to an unreasonable risk as a result of participating in this clinical trial.
15. Any clinically significant event or condition uncovered during surgery.
16. History of abuse illicit drugs, prescription medicines or alcohol within the past 2 years.
17. Known history of anti-HIV antibody positive .
18. Failure to pass drug and alcohol screen.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2014-09-21 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
the area under the curve of VAS pain intensity scores | at 1, 2, 3, 4±0.25, 8±0.5, 12±0.5, 16±0.5, 20±0.5, 24±1, 28±1, 32±2, 36±2, 40±2, 44±2, and 48±2 h after the surgery
  Pain assessment calculated as the area under the curve of VAS pain intensity scores through 48 hours

SECONDARY OUTCOMES:
Consumption of diclofenac dose | in 48 hours after surgery
  Consumption of diclofenac (Day 1-2) via Intramuscular Injection (IM injection)
Time of operation to diclofenac dose | in 48 hours after surgery
  Time from the end of operation to the first IM injection diclofenac dose
Brief Pain Inventory (BPI) | at 24h and 48h after surgery
  Brief Pain Inventory (BPI)
Patient satisfaction | at 48h after surgery
  Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Chieh Wu, MD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- General Clinical Research Center, Tri-service General Hospital, Taipei, Taiwan